CLINICAL TRIAL: NCT01198522
Title: Phase I Study of the Tumor-targeting Human L19IL2 Monoclonal Antibody-cytokine Fusion Protein in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Combination Therapy of L19IL2 and Gemcitabine in Advanced Pancreatic Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19IL2GEM-01/07; 2007-001609-81 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2022-04-15 (Actual); Status verified 2014-10

CONDITIONS: Pancreatic Cancer Patients Diagnosed With Locally Advanced or Metastatic Pancreatic Cancer Not Amenable to Curative Surgical Resection
Keywords: Interleukin, IL2, Gemcitabine, monoclonal, antibody, cytokine, tumour targeting, dose finding, fusion protein, Pancreatic cancer,; L19
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Therapy of L19IL2 and Gemcitabine (Other): Dose escalation study. Part A) Gemcitabine dose escalation. Part B) L19IL2 dose escalation.
  Interventions: Drug: L19IL2 monoclonal antibody-cytokine fusion protein in combination with gemcitabine

INTERVENTIONS:
Drug: L19IL2 monoclonal antibody-cytokine fusion protein in combination with gemcitabine — Part A) Patient cohorts will sequentially be assigned to 800 or 1,000 mg/m2 of gemcitabine. gemcitabine will be given in combination with a fixed dose of L19IL2. Part B) Patient cohorts will sequentially be assigned to 10, 15,22.5,30 or 37,5 MioIU IL2 equivalents of L19IL2. L19IL2 will be given in combination with gemcitabine at the dose recommended from Part A. Should the MTD of L19IL2 not be reached within the planned cohorts listed above, the dose of L19IL2 will be further increased following 7.5 MioIU increasing steps.
  Induction treatment: Intravenous (i.v.) infusions of L19IL2 on days 1,3,5,22,24, 26,43,45,47, followed by i.v. infusions of gemcitabine on days 1,8,15,22,29,36,43. Maintenance treatment: Patients with objective tumor responses or stable disease will receive up to 4 cycles of maintenance treatment, starting on day 57: i.v. infusions of L19IL2 on days 1 (day 57), 8,15, followed by an i.v. infusion of gemcitabine. Treatment cycles will be repeated on day 29.

SUMMARY:
Systemic treatment for advanced, non-resectable pancreatic cancer still having minimal impact on the survival of patients. Even with the application of more potent gemcitabine-based regimens, survival of more than 1 year is uncommon for advanced disease. Accordingly, there is substantial unmet needs for the improvement of treatment options. The combination and simultaneous application of tumor-targeted L19IL2 with gemcitabine could result in improved anti-cancer efficacy, based on preliminary clinical and strong preclinical data.

The primary purpose of this Phase I study is to define a safe and potentially more active treatment regimen of L19IL2 (escalating doses) combined with gemcitabine for advanced pancreatic cancer patients. Also, early signs of anticancer responses of the L19IL2/gemcitabine regimen will be assessed and compared to historical controls (gemcitabine monotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid cancer of any pathology or adenocarcinoma of the pancreas with evidence of locally advanced (non resectable Stage II or III) or metastatic disease (Stage IV).
* For advanced solid cancer patients (part A), who may have received previous chemotherapy or radiation therapy, but must be amenable for a gemcitabine treatment according to the discretion of the principal investigator.
* For pancreatic cancer patients who may have received previous chemotherapy against pancreatic cancer or local radiation for palliation if the irradiated area was not the only source of measurable or assessable disease.
* ECOG performance status ≤1.
* Patients aged >/= 18 and </= 70 years.
* Patients must have at least one uni-dimensionally measurable lesion by computed tomography as defined by RECIST V1.1 criteria. This lesion must not have been irradiated during previous treatments.
* All acute toxic effects (excluding alopecia) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v3.0) Grade ≤ 1.
* Sufficient hematologic, liver and renal function:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, haemoglobin (Hb) ≥ 9.5 g/dl.
  * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase ≤ 3 x upper limit of reference range (ULN), and total bilirubin ≤ 2.0 mg/gL unless liver involvement by the tumor, in which case the transaminase levels could be up to 5 x ULN.
  * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 50 mL/min.
* Life expectancy of at least 12 weeks.
* Documented negative test for human immunodeficiency virus.
* Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
* If of childbearing potential, agreement must be made to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* Evidence of a personally signed and dated Ethics Committee-approved Informed Consent indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

* Presence of active infections (e.g. requiring antibiotic therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Presence of known brain metastases. If patient is symptomatic, negative CT scan within two months before study beginning is required. However, presence of controlled brain metastases (i.e., evaluated as SD or PR after radiotherapy) is allowed.
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study, or any cancer curatively treated ≥ 2 yeast prior to study entry, except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumours (TA, TIs &TI).
* History of chronic hepatitis B or C, or chronic active hepatitis or active autoimmune diseases.
* History of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
* Irreversible cardiac arrhythmias requiring permanent medication.
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe rheumatoid arthritis.
* Severe diabetic retinopathy.
* History of allograft or stem cell transplantation
* Major trauma including surgery within 4 weeks of administration of study treatment.
* Known history of allergy to IL2, gemcitabine, or other intravenously administered human proteins/peptides/antibodies.
* Pregnancy or breast feeding. Female patient must agree to use effective contraception, or be surgically sterile or postmenopausal. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Chemotherapy (standard or experimental) or radiation therapy within 4 weeks of the administration of study treatment.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment.
* Patient requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion. A maximum dose per day of 5 mg prednisone (or equivalent), when it is meant to address cancer symptoms (e.g., pain, dyspnoea, lack of appetite), is allowed. A suspected presence of chronic inflammatory disease has to be considered an exclusion criterion.
* Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.
* Persons who are interned in Institutions by Judiciary or other Authorities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and the preliminary tolerability profile. | 49 days
  Establishment of the maximum tolerated dose (MTD) and the preliminary tolerability profile of L19IL2 and gemcitabine including the recommended phase II doses (RD) when used in combination.

SECONDARY OUTCOMES:
Pharmacokinetics | 4 weeks
  Investigation of the pharmacokinetics of L19IL2 and gemcitabine when given as a combination.
Human anti-fusion protein antibodies | 18 months
  Investigation of the induction of human anti-fusion protein antibodies (HAFA) levels.
Antitumor activity | 18 months
  Investigation of the antitumor activity of the combination of L19IL2 and gemcitabine in previously treated and untreated locally advanced or metastatic pancreatic cancer patients.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (2):
  - Campus Charité Virchow Klinikum, Berlin
  - National Center for Tumor Diseases (NCT), Heidelberg
- Italy (3):
  - Mater Salutis Hospital, Legnago
  - European Institute of Oncology, Milan
  - Azienda Ospedaliera Universitaria Senese, Siena